CLINICAL TRIAL: NCT03451708
Title: Optokinetic Stimulation for the Treatment of Hemispatial Neglect - Safety and Efficacy Studies
Brief Title: OKS for the Treatment of Hemispatial Neglect
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment and other trial activities were halted by COVID-19 pandemic.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Johns Hopkins University (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Chun Lim, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2016P000396; R21EY027468 (NIH)
Record Dates: First submitted 2018-02-08; First posted 2018-03-02 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Neglect, Hemispatial; Neglect, Sensory; Neglect, Hemisensory
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Optimization of OKS (Experimental): Crossover study examining various OKS protocols on improving symptoms of hemispatial neglect
  Interventions: Device: OKS
- Safety and efficacy study (Experimental): Randomized study assessing the safety and efficacy of OKS in treating hemispatial neglect
  Interventions: Device: OKS
- Effect of repetitive stimulation (Experimental): Benefits of daily, repetitive OKS in treating hemispatial neglect
  Interventions: Device: OKS
- OKS and gait (Experimental): Effect of OKS on gait and balance
  Interventions: Device: OKS

INTERVENTIONS:
Device: OKS — Optokinetic stimulation will be displayed on a see-through liquid crystal display lens placed in front of the subjects.

SUMMARY:
Hemispatial neglect is a disorder where the patient has difficulty attending to objects and information in the left side of space, which occurs following strokes to the right side of the brain. This project is designed to help us understand how optokinetic stimulation treats the symptoms of hemispatial neglect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with right hemispheric lesions resulting in hemispatial neglect as confirmed by Behavioral Inattention Test or Center of Cancellation Test

Exclusion Criteria:

* Reduced vision
* Documented vestibular disorder

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Hemispatial neglect scores | After 1 hour of OKS
  Performance on Center of Cancellation Test
Change in Hemispatial neglect scores | After 1 hour of OKS
  Performance on Behavioral Inattention Test
Effect of OKS on vision | After 1 hour of OKS
  visual acuity
Effect of OKS on vision | After 1 hour of OKS
  reading speed

SECONDARY OUTCOMES:
Changes in secondary hemispatial neglect scores | After 1 hour of OKS
  Line bisection score
Changes in secondary hemispatial neglect scores | After 1 hour of OKS
  grip strength
Changes in secondary hemispatial neglect scores | After 1 hour of OKS
  extinction score
Effect of OKS on gait | After 1 hour of OKS
  Gait assessment
Effect of OKS on gait | After 1 hour of OKS
  Balance assessments

CONTACTS AND LOCATIONS:
Overall Officials: Chun Lim, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963